CLINICAL TRIAL: NCT04709055
Title: Implementation of coMplex PeRi-OperatiVe intervEntion in olDer Patients With Cancer : a Multicenter Randomized Controlled Trial
Brief Title: Complex Peri-operative Intervention in Older Patients With Cancer
Acronym: IMPROVED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Société Francophone d'Onco-Gériatrie (Other); Federation of Research in Surgery (FRENCH) (Other); PACAN - Plateforme de Recherche Clinique Patients Agés et Cancer (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: APHP180675; 2020-A01354-35 (Other: N° IDRCB)
Record Dates: First submitted 2020-10-28; First posted 2021-01-14 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2020-09

CONDITIONS: Digestive Cancer
Keywords: Age; Geriatric Assesment; Co-management; Surgery; Digestive Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Co-management arm (geriatric and surgical) (Experimental)
  Interventions: Other: Co-management
- Usual care (Active Comparator)
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Co-management — Personalized and intensive geriatric peri-operative care
  Arms: Co-management arm (geriatric and surgical)
Other: Usual care — Pre-operative and post-operative geriatric care as per usual practice
  Arms: Usual care

SUMMARY:
Incidence of digestive cancers increase and half of new cases will be people of 75 years or more in 2050. Surgery is one of the main treatment's strategy but post-operative morbi-mortality increases with age. Pre-operative Geriatric Assessment enable to identify frail or vulnerable patients at risk of post-operative complications.

The coordinating team postulate that a geriatric and surgical co-management with a combination of several targeted geriatric interventions with usual post-operative care could improve the post-operative care and decrease the risk of morbi-mortality in older patients with digestive cancers.

DETAILED DESCRIPTION:
Multicenter Randomized Clinical Trial in 2 parallel-groups with masked adjudication of main endpoint

ELIGIBILITY:
Inclusion Criteria:

* Aged 75 years or more
* Gastric, colo-rectal, pancreatic cancer or hepatic metastasis needed a surgical treatment
* Health Insurance
* At risk of post-operative complication through Surgical Risk Calculator (>25%) or surgeon judgment.
* Written consent

Exclusion Criteria:

* Surgery in emergency

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 630 (Estimated)
Dates: Start 2021-01-14 (Estimated); Primary Completion 2024-08-14 (Estimated); Study Completion 2024-10-14 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with postoperative complications of grade II or higher in the Clavien-Dindo | at 30 days after surgery

SECONDARY OUTCOMES:
Percentage of patients with postoperative complications of each grade in the Clavien-Dindo | at Day 14 and Day 30
Percentage of patients with each complication among a prespecified list of complication | at Day 14 and Day 30
Social Status | at Day 14 and Day 30 after surgery
Activities of Daily Living Scale | at Day 14 and Day 30 after surgery
Instrumental Activities of Daily Living Scale | at Day 14 and Day 30 after surgery
Mini-Geriatric Depressive Scale | at Day 14 and Day 30 after surgery
Mini cognitive scale | at Day 14 and Day 30 after surgery
Updated Charlson Comorbidity Index | at Day 14 and Day 30 after surgery
Mini Nutritional Assessment-Short Form | at Day 14 and Day 30 after surgery
Body mass index | at Day 14 and Day 30 after surgery
Timed Up and Go | at Day 14 and Day 30 after surgery
Gait speed | at Day 14 and Day 30 after surgery
Percentage of patients with cancelled surgeries | at Day 0 to Day 8
Percentage of patients with postponed surgeries | at Day 0 to Day 8
Percentage of patients with complete intervention in the experimental arm | at Day 0 to Day 8
Time of onset of each post-operative complication | at Day 14, Day 30 and Day 90 after surgery
Percentage of patients transfered to geriatric unit, intensive care unit, rehabilitation unit or other departement. | at Day 14, Day 30 and Day 90 after surgery
Length of stay to geriatric unit, intensive care unit, rehabilitation unit or other departement. | at Day 14, Day 30 and Day 90 after surgery
Quality of life (European Organisation for Research and Treatment of Cancer - Quality of life - C30) | at Day 30 and Day 90 after surgery
Quality of life (European Organisation for Research and Treatment of Cancer - Quality of life - ELD14) | at Day 30 and Day 90 after surgery
Overall survival | at Day 30 and Day 90 after surgery
Length of hospitalizations | at Day 14 after surgery
Percentage of patients returned at home or institutionalization | at Day 14, Day 30 and Day 90 after surgery
Autonomy (Activities of Daily Living scale) | at Day 14 , Day 30 and Day 90 after surgery
Patient and professionals experience (ancillary study using semi-directive interviews) | at Day 30 after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Elena PAILLAUD LAURENT PUIG, MD, PhD, Principal Investigator — Assistance Publique Hôpitaux de Paris (AP-HP)
Locations (1):
- Assistance Publique Hôpitaux de Paris - Hôpital européen Georges-Pompidou, Paris, France